CLINICAL TRIAL: NCT05872100
Title: THE EFFECT OF MINDFULNESS-BASED PRACTICES GIVEN TO NURSING STUDENTS ON COMPASSION, COMPASSION AND NURSING CARE
Brief Title: THE EFFECT OF MINDFULNESS-BASED PRACTICES GIVEN TO NURSING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tuğba Bilgehan (Other)
Responsible Party: Sponsor-Investigator, Tuğba Bilgehan, Asst Prof, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TUGBABILGEHAN
Record Dates: First submitted 2023-04-25; First posted 2023-05-24 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Nurse's Role
Keywords: mindfulness; nursing; awareness; nursing care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RESPONSE GROUP (Experimental): Mindfulness-based psycho-education program will be applied to the students in the experimental group. After the end of the study, the mindfulness-based psychoeducation program given in the experimental group will also be applied to the control group. A 45-minute training and preliminary information will be given to the student group. Participants will meet for the first session. After the trainer, who is a clinical psychologist, introduces himself and meets the participants, 10 minutes will be given to ensure that all participants meet and look at each other. Then, the aim of the research will be discussed by sharing the content of the three-week program. After three weeks, post-tests will be administered.
  Interventions: Behavioral: MINDFULNESS BASED APPLICATION
- control group (No Intervention): A pre-test will be applied to the control group. No intervention will be made. The final test will be applied.

INTERVENTIONS:
Behavioral: MINDFULNESS BASED APPLICATION — * The effectiveness of mindfulness practices in the field of health
  * Breathing exercise
  * Discussing and sharing about exercise
  * Introduction of informal and formal mindfulness practices
  * Communication exercise with conscious awareness
  * Sounds and thoughts meditation
  * The concept of compassion
  * Biological foundations of compassion
  * Self-compassion
  * Barriers to compassion
  * Coping with compelling emotions
  * Coping with the intensity of compassion
  * Compassionate mindfulness attitudes
  * Admission stages and improving acceptance
  * Compassion Meditation
  * Courtesy Meditation
  * My partner activity
  * Body Scan
  * Mindfulness Sitting Meditation
  * Receiving feedback on the development of mindfulness skills and the content of the training program
  * Integration of conscious awareness exercises in daily life for the future
  Arms: RESPONSE GROUP

SUMMARY:
In our research, it is expected that the 'conscious awareness-based psychoeducation program' will be made to the nursing students who go into clinical practice, to increase the level of mindfulness of the students, to increase their level of compassion and compassion, and to reflect this awareness while providing nursing care. It is thought that it is important to evaluate the effects of mindfulness-based psychoeducation program practices on nursing care and to evaluate mindfulness-based psychoeducation program practices.

This study was planned as a randomized control study with an intervention group to determine the effect of mindfulness-based practices given to nursing students on compassion, compassion and nursing care.

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years old
* become a nursing student
* Having successfully passed the internal medicine nursing course

Exclusion Criteria:

* not attending 1 session of the study
* unwillingness to quit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
THE EFFECT OF MINDFULNESS-BASED PRACTICES GIVEN TO NURSING STUDENTS ON COMPASSION, COMPASSION AND NURSING CARE Compassion and Compassion | 1 month
  Compassion and Compassion Scale: Developed by Hakan and Nusret (2019), 5-point Likert type (1) Not true for me at all, (2) Not true for me, (3) Neither true nor false, (4) True for me and (5) The scale, which is very correct for me, consists of 15 items. The scale consists of 3 sub-dimensions, self-centeredness, compassion and compassion. Increasing scores indicate an increase in the value of the relevant dimension. The score that can be obtained from the scale ranges from 15-75. Caring Behaviors Scale: This scale, created by Wu et al. (2006), is an abbreviated form of the 42-item "Caring Behaviors Scale-42" developed by Wolf et al. (1994) and suitable for bilateral diagnosis by patients and nurses (12). The current form of the scale is designed in a 6-point Likert type consisting of 24 questions and measures the care behaviors of healthcare workers.
THE EFFECT OF MINDFULNESS-BASED PRACTICES GIVEN TO NURSING STUDENTS ON COMPASSION, COMPASSION AND NURSING CARE Caring Behaviors | 1 month
  Caring Behaviors Scale: This scale, created by Wu et al. (2006), is an abbreviated form of the 42-item "Caring Behaviors Scale-42" developed by Wolf et al. (1994) and suitable for bilateral diagnosis by patients and nurses (12). The current form of the scale is designed in a 6-point Likert type consisting of 24 questions and measures the care behaviors of healthcare workers.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Bilgehan, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No